CLINICAL TRIAL: NCT01563237
Title: Safety and Performance of Miami InnFocus Drainage Implant (MIDI Arrow) to Relieve Glaucoma Symptoms
Brief Title: Safety and Performance of Miami InnFocus Drainage Implant (MIDI Arrow) Glaucoma Drainage Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnFocus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN004
Record Dates: First submitted 2012-03-21; First posted 2012-03-26 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIDI Arrow (Experimental): Implantation of MIDI Arrow
  Interventions: Device: MIDI Arrow

INTERVENTIONS:
Device: MIDI Arrow — Implantation of MIDI Arrow
  Other Names: Glaucoma drainage device implantation

SUMMARY:
To assess the safety and performance of the MIDI Arrow in patients suffering from glaucoma that is inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥ 18 mm Hg and ≤ 40 mm Hg

DETAILED DESCRIPTION:
This will be a monocentric, non-randomized, single arm clinical study in which each patient meeting the inclusion criteria and not excluded per the exclusion criteria will be implanted with a MIDI Arrow in the anterior chamber of the eye. Patients will be followed for at least 24 months with an expected enrollment period of up to 24 months. Safety of the shunt will be evaluated with indirect and direct microscopic evaluation of the implanted and non-implanted eyes pre and post operatively, and at defined follow-up intervals for hypotony, inflammation, infection, migration of the shunt, visual acuity, as well as a number of other defined potential complications. The effectiveness of the shunt will be evaluated by measurement of intraocular pressure at defined intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, age 18 to 85 years, inclusive
2. Patient has primary open angle glaucoma that is inadequately controlled on tolerated medical therapy with intraocular pressure greater than or equal to 18 mm Hg and less than or equal to 40 mm Hg
3. Patient must have signed and dated the Informed Consent form

Exclusion Criteria:

1. Unwilling or unable to give informed consent or unable to return for scheduled protocol visits.
2. Pregnant or nursing women.
3. No light perception.
4. Active iris neovascularization or active proliferative retinopathy.
5. Iridocorneal endothelial syndrome.
6. Epithelial or fibrous downgrowth.
7. Pseudoexfoliative glaucoma
8. Aphakia.
9. Vitreous in anterior chamber for which a vitrectomy is anticipated.
10. Corneal disease
11. Acute, chronic or recurrent uveitis.
12. Severe posterior blepharitis.
13. Unwilling to discontinue contact lens use after surgery.
14. Previous ophthalmic surgery, excluding phacoemulsification (cataract) surgery or corneal refractive surgery.
15. Prior cataract surgery involving a conjunctival incision
16. Need for glaucoma surgery combined with other ocular procedures except for cataract surgery or anticipated need for additional ocular surgery during the investigational period.
17. Less than 0.1 (20/200) visual acuity in the non-test eye.
18. Infectious conjunctivitis, a narrow-angle glaucoma, endophthalmitis, orbital cellulitis one, infection, severe dry eye, severe myopia, conjunctivitis fine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-06; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle M Riss, MD, Principal Investigator — Clinique Mutualiste de Pessac, Pessac, France
Locations (1):
- Clinique Mutualiste - Pavillon Ophtalmogique, Pessac, France

REFERENCES:
- [Derived] Garcia-Feijoo J, Batlle JF, Aptel F, Lachkar Y, Riss I, Sadruddin O, Nguyen T, Beckers HJM. Pooled Analysis of Three MicroShunt Studies in Primary Open-Angle Glaucoma Evaluating Different Concentrations of Applied Mitomycin C. Ophthalmol Ther. 2025 Jul;14(7):1533-1549. doi: 10.1007/s40123-025-01149-4. Epub 2025 May 23. PMID 40408035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Listing of Eyes under Study
Units Other Than Participants: Eyes
Groups:
- First Studied Eye; Second Studied Eye: Patients suffering from glaucoma that is inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥ 18 mm Hg and ≤ 40 mm Hg.
Period: Overall Study
Arm/Group | First Studied Eye | Second Studied Eye
Started (69 Participants and 74 eyes were enrolled) | 64; 69 Eyes | 5; 5 Eyes
Completed (59 participants and 64 eyes completed the study) | 54; 59 Eyes | 5; 5 Eyes
Not Completed | 10; 10 Eyes | 0; 0 Eyes
Not completed — Lost to Follow-up | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Medical Reasons | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all enrolled subject who have signed the informed consent and attended the procedure visit to receive the assigned therapy under evaluation (MIDI Arrow).
Groups:
- MIDI Arrow: Implantation of MIDI Arrow (MicroShunt) in the anterior chamber of the eye in patients with primary open angle glaucoma (POAG)
Arm/Group | MIDI Arrow
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 39
Region of Enrollment [Count of Participants; unit: Participants]
  France | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes With Study Success
Description: The rate of success reflected sustained control of IOP over 24 Months from baseline
Time Frame: Months 6, 9, 12 and 24
Population: The Intent-to-Treat (ITT) population included all enrolled eyes who have signed the informed consent and attended the procedure visit to receive the assigned therapy under evaluation (MIDI Arrow).
Measure: Count of Units; unit: Implanted eyes
Units Other Than Participants: Implanted eyes
Groups:
- Success With Respect to IOP: The rates of success reflected sustained control of IOP
Arm/Group | Success With Respect to IOP
Number analyzed (Participants) | 67
Number analyzed (Implanted eyes) | 72
Implanted eyes
  Month 6 | 50
  Month 9 | 52
  Month 12 | 50
  Month 24 | 51

2. Secondary Outcome: IOP Change From Baseline
Description: Intraocular Pressure (IOP) change in studied eye compared to baseline value at all timepoints thru 24 Months.
Time Frame: At Day 1, Day 7, Week 3, Week 6, Month 3, Month 9, Month 12 and Month 24
Population: The Intent-to-Treat (ITT) population included all enrolled subject who have signed the informed consent and attended the procedure visit to receive the assigned therapy under evaluation (MIDI Arrow).
  IOP data collected after glaucoma re-operation was censored for this analysis
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Groups:
- IOP Change From Baseline: Change of IOP relative to the pre-operative value
Arm/Group | IOP Change From Baseline
Number analyzed (Participants) | 67
Number analyzed (eyes) | 72
mmHg
  IOP at Baseline | 26 (7)
  Day 1: number analyzed (eyes) | 69
  Day 1 | 9.2 (4.2)
  Day 7: number analyzed (eyes) | 70
  Day 7 | 10.9 (5.2)
  Week 3: number analyzed (eyes) | 69
  Week 3 | 13.2 (6.3)
  Week 6: number analyzed (eyes) | 67
  Week 6 | 13.3 (5.2)
  Month 3: number analyzed (eyes) | 68
  Month 3 | 13.8 (4.1)
  Month 6: number analyzed (eyes) | 68
  Month 6 | 15 (3.9)
  Month 9: number analyzed (eyes) | 66
  Month 9 | 15.4 (4.2)
  Month 12: number analyzed (eyes) | 67
  Month 12 | 15.6 (4.7)
  Month 24: number analyzed (eyes) | 61
  Month 24 | 16.2 (5.8)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported for the duration of the study of 24 Months.
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) affecting the study eye. Adverse Events were collected and reported per eye.
Groups:
- Study Eyes Selected to be Operated Within the Study: Patients suffering from glaucoma that is inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥ 18 mm Hg and ≤ 40 mm Hg.
Arm/Group | Study Eyes Selected to be Operated Within the Study
All-Cause Mortality (participants affected / at risk) | 1/74
Serious Adverse Events (participants affected / at risk) | 10/74
Other Adverse Events (participants affected / at risk) | 68/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Eyes Selected to be Operated Within the Study (N=74)
Intraocular Pressure Increased (Investigations) | 3 (3)
Gallbladder Operation (Surgical and medical procedures) | 1 (1)
Medical Device Repositioning (Surgical and medical procedures) | 1 (1)
Macular Degeneration (Eye disorders) | 1 (1)
Macular Oedema (Eye disorders) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 1 (1)
Conjunctival Filtering Bleb Leak (Injury, poisoning and procedural complications) | 1 (1)
Perforation Bile Duct (Hepatobiliary disorders) | 1 (1)
Dacryocystitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Eyes Selected to be Operated Within the Study (N=74)
Intraocular pressure increased (Investigations) | 39 (64)
Hyphaema (Eye disorders) | 19 (19)
Hypotony of eye (Eye disorders) | 13 (15)
Cataract (Eye disorders) | 17 (17)
Macular oedema (Eye disorders) | 3 (6)
Diplopia (Eye disorders) | 2 (2)
Keratitis (Eye disorders) | 12 (12)
Visual acuity reduced (Eye disorders) | 4 (6)
Eye irritation (Eye disorders) | 5 (6)
Ulcerative keratitis (Eye disorders) | 5 (6)
Eyelid ptosis (Eye disorders) | 4 (4)
Conjunctival haemorrhage (Eye disorders) | 2 (2)
Iris adhesions (Eye disorders) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Retinopathy (Eye disorders) | 2 (2)
Eyelid irritation (Eye disorders) | 1 (2)
Allergic Keratitis (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Blepharospasm (Eye disorders) | 1 (1)
Choroidal detachment (Eye disorders) | 1 (1)
Corneal irritation (Eye disorders) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1)
Eye Haemorrhage (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Lacrimal Disorder (Eye disorders) | 1 (1)
Macular Degeneration (Eye disorders) | 1 (1)
Narrow Anterior Chamber Angle (Eye disorders) | 1 (1)
Trichiasis (Eye disorders) | 1 (1)
Intraocular Pressure Decreased (Investigations) | 2 (2)
Drug Intolerance (General disorders) | 7 (7)
Conjunctival Abrasion (Injury, poisoning and procedural complications) | 1 (1)
Conjunctival Filtering Bleb Leak (Injury, poisoning and procedural complications) | 1 (1)
Conjunctival Scar (Injury, poisoning and procedural complications) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 1 (1)
Conjunctivitis (Infections and infestations) | 3 (3)
Dacryocystitis (Infections and infestations) | 1 (2)
Infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Visual Field Defect (Nervous system disorders) | 2 (2)
Device Deployment Issue (Product Issues) | 3 (3)
Device Difficult To Use (Product Issues) | 1 (1)
Device Occlusion (Product Issues) | 1 (1)
Gallbladder Operation (Surgical and medical procedures) | 1 (1)
Medical Device Repositioning (Surgical and medical procedures) | 1 (1)
Suture Removal (Surgical and medical procedures) | 1 (1)
Perforation Bile Duct (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes